CLINICAL TRIAL: NCT00448552
Title: Treatment of Relapsed or Metastatic Head and Neck Carcinomas With Oxaliplatin and Capecitabine
Brief Title: Oxaliplatin and Capecitabine in Treating Patients With Relapsed or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: 20030243; SCCC-2003050 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20060071 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage IV salivary gland cancer; untreated metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving oxaliplatin together with capecitabine works in treating patients with relapsed or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with chemotherapy naïve relapsed or metastatic head and neck cancer treated with oxaliplatin and capecitabine.

Secondary

* Evaluate the safety and toxicity of this regimen in these patients.
* Determine the one-year survival and overall survival of these patients.

OUTLINE: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 2-15. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed head and neck cancer

  * Relapsed or metastatic disease
* Measurable disease
* No CNS metastases (unless CNS metastases have been stable for > 3 months)
* No clinically significant pericardial effusion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Absolute granulocyte count > 1,500/mm³
* Platelet count > 100,000/mm³
* Bilirubin < 2.0 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Alkaline phosphatase < 2.5 times ULN (5 times ULN if liver metastases are present or 10 times ULN if bone disease is present)
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No clinically serious, uncontrolled cardiovascular disease
* No New York Heart Association class III-IV heart disease
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No unstable angina
* No arrhythmia
* No concurrent serious, uncontrolled infections
* No other cancer requiring treatment within the past 5 years, except cured nonmelanoma skin cancer or treated in situ cervical cancer
* No loss of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* No history of persistent neurosensory disorder including, but not limited to, peripheral neuropathy
* No history of uncontrolled seizures or CNS disorders
* No history of psychiatric disability or other serious uncontrolled medical condition that would preclude study compliance
* No history of clinically significant interstitial lung disease and/or pulmonary fibrosis
* No prior hypersensitivity or unanticipated severe reaction to fluoropyrimidine therapy, fluorouracil, or platinum-based compounds

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic or relapsed disease
* More than 4 weeks since prior major surgery and recovered
* More than 4 weeks since prior participation in any investigational drug study
* At least 6 months since prior adjuvant fluoropyrimidine therapy

  * No other prior fluoropyrimidines
* At least 6 months since prior adjuvant platinum-based therapy

  * No other prior platinum-based therapy
* No concurrent radiotherapy to the head and neck
* No other concurrent chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-04 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete response and partial response)

SECONDARY OUTCOMES:
Toxicity as measured by NCI CTC
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Luis E. Raez, MD, FACP, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States